CLINICAL TRIAL: NCT04629248
Title: A Phase III Randomized, Open-Label Active Comparator-Controlled Multicenter Study to Evaluate Efficacy and Safety of Obinutuzumab in Patients With Primary Membranous Nephropathy
Brief Title: A Study Evaluating the Efficacy and Safety of Obinutuzumab in Participants With Primary Membranous Nephropathy
Acronym: MAJESTY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WA41937; 2020-003233-38 (EudraCT Number); 2023-506525-11-00 (Other: EU CT Number)
Record Dates: First submitted 2020-10-27; First posted 2020-11-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Primary Membranous Nephropathy
MeSH Terms: interventions — obinutuzumab; Tacrolimus; Methylprednisolone; Acetaminophen; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Open Label Treatment: Obinutuzumab (Experimental): Participants will be randomized at a 1:1 ratio to receive open-label treatment with obinutuzumab according to region and anti-phospholipase A2 receptor (PLA2R) autoantibody titer (using Euroimmun ELISA).
  Interventions: Drug: Obinutuzumab; Drug: Methylprednisolone; Drug: Acetaminophen; Drug: Diphenhydramine
- Open Label Treatment: Tacrolimus (Active Comparator): Participants will be randomized at a 1:1 ratio to receive open-label treatment with tacrolimus according to region and anti-PLA2R autoantibody titer (using Euroimmun ELISA).
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Obinutuzumab — Open Label: An intravenous (IV) infusion of 1000 milligram (mg) of obinutuzumab will be administered at Week 0, Week 2, Week 24, and Week 26. Participants who relapse during the open-label treatment period may be eligible for further treatment.
  Other Names: Gazyva
  Arms: Open Label Treatment: Obinutuzumab
Drug: Tacrolimus — Open Label: Participants will receive tacrolimus at a starting oral dose (PO) of 0.05 mg/kilogram (kg) (participant dry weight) per day divided into two equal doses given at 12-hour intervals, titrated to serum trough level 5-7 Nanograms per millilitre (ng/mL). Optimized tacrolimus dose will be maintained for a maximum 52 weeks dependent on response and then tapered over 8 weeks. Participants who relapse during the open-label treatment period will have their dose of tacrolimus tapered over 8 weeks and may be eligible for further treatment.
  Arms: Open Label Treatment: Tacrolimus
Drug: Methylprednisolone — Premedication: Methylprednisolone 80 mg IV will be administered between 30 and 60 minutes prior to the obinutuzumab infusion in all study periods.
  Arms: Open Label Treatment: Obinutuzumab
Drug: Acetaminophen — Premedication: Acetaminophen (650-1000 mg, or equivalent dose of a similar agent) PO or IV will be administered between 30 and 60 minutes prior to the obinutuzumab infusion in all study periods.
  Arms: Open Label Treatment: Obinutuzumab
Drug: Diphenhydramine — Premedication: Diphenhydramine (50 mg, or equivalent dose of a similar agent) PO or IV will be administered between 30 and 60 minutes prior to the obinutuzumab infusion in all study periods.
  Arms: Open Label Treatment: Obinutuzumab

SUMMARY:
This study will evaluate the efficacy, safety, pharmacodynamics, and pharmacokinetics (PK) of obinutuzumab compared with tacrolimus in participants with primary membranous nephropathy (pMN).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary membranous nephropathy (pMN) according to renal biopsy prior to or during screening
* Screening urinary protein-to-creatinine ratio (UPCR) >= 5 g/g from 24-hour urine collection after best supportive care for >= 3 months prior to screening or screening UPCR >= 4 g/g after best supportive care for >= 6 months prior to screening
* eGFR >= 40 mL/min/1.73m^2 or qualified endogenous creatinine clearance >= 40 mL/min/1.73m^2 based on 24-hour urine collection during screening
* Other inclusion criteria may apply

Exclusion Criteria:

* Participants with a secondary cause of MN
* Pregnancy or breastfeeding
* Evidence of >= 50% reduction in proteinuria during the previous 6 months prior to randomization
* Severe renal impairment, including the need for dialysis or renal replacement therapy
* Type 1 or 2 diabetes mellitus
* Receipt of an excluded therapy, including any anti-CD20 therapy less than 9 months prior to or during screening; or cyclophosphamide, tacrolimus, or cyclosporin less than 6 months prior to or during screening
* Significant or uncontrolled medical disease which, in the investigator's opinion, would preclude participant participation
* Known active infection of any kind or recent major episode of infection
* Major surgery requiring hospitalization within the 4 weeks prior to screening
* Current active alcohol or drug abuse or history of alcohol or drug abuse within 12 months prior to screening
* Intolerance or contraindication to study therapies
* Other exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2027-12-21 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve a Complete Remission (CR) at Week 104 | Week 104

SECONDARY OUTCOMES:
Percentage of Participants who Achieve an Overall Remission at Week 104 | Week 104
Percentage of Participants who Achieve CR at Week 76 | Week 76
Time to Treatment Failure, Meeting Escape Criteria, or Relapse after Complete or Partial Remission | Up to 8 years
Time to a Sustained Reduction of Estimated Glomerular Filtration Rate (eGFR) >= 30% from Baseline | Up to 8 years
Mean Change in T-score from Baseline in the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Scale at Week 104 | Baseline to Week 104
  Self-reported changes in fatigue will be measured using the PROMIS Fatigue Scale.
Duration of CR | Up to 8 years
Change in anti-PLA2R Autoantibody Titer | Baseline to Week 52
Mean Change from Baseline in the PROMIS Global Assessment of Physical Health Scale at Week 104 | Baseline to Week 104
  Self-reported changes in physical health will be measured using the PROMIS Physical Health Scale
Percentage of Participants with Adverse Events (AEs) | Up to 8 years
  Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Percentage of Participants with AEs of Special Interest (AESIs) | Up to 8 years
  AESIs are required to be reported by the investigator to the Sponsor immediately
Peripheral B-cell Counts at Specified Timepoints | Weeks 0 (baseline), 2, 4, 12, 24, 26, 36, 52, 64, 76, 88, 104, 117, 130, 156, 182, 208 and every 26 weeks thereafter
Serum Concentrations of Obinutuzumab at Specified Timepoints | Weeks 0 (baseline), 2, 4, 12, 24, 26, 36, 52, 64, 76, 88, 104, 117, 130, 143, 156, 169, 182, 195, 208, every 26 weeks thereafter
Prevalence of Anti-drug Antibodies (ADAs) to Obinutuzumab at Baseline | Open Label: Baseline; Escape Treatment: Week 0
Incidence of ADAs during the study | Weeks 2, 4, 12, 24, 26, 36, 52, 64, 76, 88, 104, 130, 156, 182, 208 and every 26 weeks thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (50):
- United States (8):
  - Kaiser Permanente - San Francisco Medical Center, San Francisco, California
  - University of Colorado in Denver-Anschutz Medical Campus, Aurora, Colorado
  - Accel Research Sites; Mid-Florida Kidney and Hypertension Care, Altamonte Springs, Florida
  - University of Iowa, Iowa City, Iowa
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - Nephrotex Research Group, Dallas, Texas
- Argentina (3):
  - Organizacion Medica de Investigacion, Buenos Aires
  - CINME, Buenos Aires
  - Hospital Britanico Buenos Aires, Buenos Aires
- Brazil (4):
  - Ser Servicos Especializados Em Reumatologia, Salvador, Estado de Bahia
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital do Rim e Hipertensão - Fundação Oswaldo Ramos, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
- China (10):
  - Zhejiang Provincial People?s Hospital, Hangzhou, Zhejiang
  - Peking University First Hospital, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - The 1st Affiliated hospital of Fujian Medical University, Fuzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Huashan Hospital, Fudan University, Shanghai
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xian Jiao Tong University, Xi'an
  - General Hospital of Ningxia Medical University, Yinchuan
- France (3):
  - Hopital Henri Mondor, Créteil
  - Hopital Tenon, Paris
  - Hopital Rangueil, Toulouse
- Sheba MC, Ramat Gan, Israel
- Italy (5):
  - Policlinico di Bari, Bari, Apulia
  - A.O. U. Federico II, Napoli, Campania
  - A.O. Spedali Civili Di Brescia-P.O. Spedali Civili, Brescia, Lombardy
  - ASST Monza - Ospedale San Gerardo, Monza, Lombardy
  - Ospedale San Giovanni Bosco, Turin, Piedmont
- Poland (5):
  - Uniwersytecki Szpital Kliniczny nr 1 im. N. Barlickiego, ?ód?
  - Uniwersytecki Szpital Kliniczny im WAM CSW, ?ód?
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bia?ystok
  - Szpital Uniwersytecki im.dr.A.Jurasza w Bydgoszczy, Bydgoszcz
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroc?aw
- Russia (3):
  - First Moscow State Medical University n.a. I.M. Sechenov, Moscow, Moscow Oblast
  - Rostov State Medical Uni, Rostov-on-Don, Rostov Oblast
  - German clinic, Saint Petersburg, Sankt-Peterburg
- Spain (5):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Turkey (Türkiye) (3):
  - Hacettepe Uni School of Medicine, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Ege Uni School of Medicine, Izmir

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Dossier C, Bonneric S, Baudouin V, Kwon T, Prim B, Cambier A, Couderc A, Moreau C, Deschenes G, Hogan J. Obinutuzumab in Frequently Relapsing and Steroid-Dependent Nephrotic Syndrome in Children. Clin J Am Soc Nephrol. 2023 Dec 1;18(12):1555-1562. doi: 10.2215/CJN.0000000000000288. Epub 2023 Sep 6. PMID 37678236
- [Derived] Dossier C, Hogan J. Response to Majeranowski. Pediatr Nephrol. 2021 Jun;36(6):1653. doi: 10.1007/s00467-021-04982-4. Epub 2021 Mar 10. No abstract available. PMID 33693991